CLINICAL TRIAL: NCT03222427
Title: An Absolute Bioavailability Study of LY3314814 in Healthy Subjects Using an Intravenous Tracer Method
Brief Title: A Study of LY3314814 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15993; I8D-MC-AZEP (Other: Eli Lilly and Company.); 2017-001181-18 (EudraCT Number)
Record Dates: First submitted 2017-07-18; First posted 2017-07-19 (Actual); Results first posted 2019-03-22 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Healthy

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3314814 (Experimental): Single 50 milligram (mg) dose of LY3314814 administered orally
  Interventions: Drug: LY3314814
- [13C415N3] LY3314814 (Experimental): Single 100 micrograms (μg) intravenous (IV) dose of [13C415N3] LY3314814 administered as an IV infusion.
  Interventions: Drug: [13C415N3] LY3314814

INTERVENTIONS:
Drug: LY3314814 — Administered orally
  Arms: LY3314814
Drug: [13C415N3] LY3314814 — Administered as an IV infusion
  Arms: [13C415N3] LY3314814

SUMMARY:
The purpose of this study is to measure how much LY3314814 gets into the bloodstream when it is given as a single dose by mouth and as an intravenous (IV) infusion over two hours. The study will last at least two weeks for each participant, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females
* Have venous access sufficient to allow for blood sampling and intravenous (IV) administration of the investigational product

Exclusion Criteria:

* Have a history of significant ophthalmic disease
* Have vitiligo or any other clinically significant disorder of skin pigmentation
* Have a history of use of antipsychotic drugs, or chronic use of antidepressant or anxiolytic drugs, prescribed as well as non-prescribed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Leeds, West Yorkshire, United Kingdom

REFERENCES:
- See also: CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=15993&attachmentIdentifier=d26671aa-b544-49ec-a1e9-9d1f5824e662&fileName=CSP_NCT03222427.pdf&versionIdentifier=
- See also: SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=15993&attachmentIdentifier=ee4534f9-f2b8-40d5-850d-11d1f36815df&fileName=SAP_NCT03222427.pdf&versionIdentifier=
- See also: CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=15993&attachmentIdentifier=7340dd9d-6193-43c0-a5eb-2df1fd900417&fileName=CSP_NCT03222427.pdf&versionIdentifier=
- See also: SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=15993&attachmentIdentifier=b5a87be9-3005-4b1b-af5b-2c213273e40a&fileName=SAP_NCT03222427.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- LY3314814 + [13C415N3] LY3314814: Single 50 milligram (mg) dose of LY3314814 administered orally simultaneously with a single 100 microgram (μg) intravenous (IV) infusion of [13C415N3] LY3314814 over 2 hours on Day 1.
Period: Overall Study
Arm/Group | LY3314814 + [13C415N3] LY3314814
Started | 8
Received One Dose of Study Drug | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug.
Arm/Group | LY3314814 + [13C415N3] LY3314814
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 8

OUTCOME MEASURES:

1. Primary Outcome: Absolute Bioavailability of LY3314814
Description: Absolute bioavailability was quantified using a mixed-effects analysis of variance (ANOVA) model applied to the log-transformed dose-normalized AUC(0-∞) of LY3314814 oral dosing and IV administered [13C415N3]-LY3314814.
Time Frame: Day 1: Predose:0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24, 48, 72, 96 and 120 hours post-dose
Population: All participants who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter per mg
Groups:
- LY3314814: Single 50 mg dose of LY3314814 administered orally.
- [13C415N3] LY3314814: Single 100 μg IV dose of [13C415N3] LY3314814 administered as an IV infusion.
Arm/Group | LY3314814 | [13C415N3] LY3314814
Number analyzed (Participants) | 8 | 7
nanogram*hour per milliliter per mg | 60.5 (41) | 59.2 (17)
Statistical Analysis 1: Comparison: LY3314814 vs [13C415N3] LY3314814; Test type: Other; Ratio of Geometric Least Squares Means = 0.952, 90% CI 2-sided [0.769 to 1.18]

2. Secondary Outcome: Pharmacokinetics: Area Under the Drug Concentration-Time Curve From Zero to Infinity (AUC[0 ∞]) of LY3314814 and [13C415N3] LY3314814
Description: Pharmacokinetics: Area Under the Drug Concentration-Time Curve from Zero to Infinity (AUC[0 ∞]) of LY3314814 and [13C415N3] LY3314814
Time Frame: Day 1: Predose:0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 24, 48, 72, 96 and 120 hours post-dose
Population: All participants who received one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | LY3314814 | [13C415N3] LY3314814
Number analyzed (Participants) | 8 | 7
nanogram*hour per milliliter (ng*hr/mL) | 3020 (41) | 5.92 (17)

ADVERSE EVENTS:
Time Frame: From baseline to end of study (Up To 7 days)
Description: All participants who have received at least one dose of study drug.
Arm/Group | LY3314814 + [13C415N3] LY3314814
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3314814 + [13C415N3] LY3314814 (N=8)
Nasopharyngitis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/27/NCT03222427/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT03222427/SAP_001.pdf